CLINICAL TRIAL: NCT05079633
Title: A Parallel Group, Prospective, Randomized, Double-blind, Two-arm, Single-center Study to Evaluate the Immunogenicity, Safety, and Tolerability of mRNA-1273 in Heterologous Prime-Boost With MVC-COV1901 in Adult Volunteers of 20 to 70 Years
Brief Title: A Heterologous Prime-boost Study to Evaluate Immunogenicity and Safety of mRNA-1273 With MVC-COV1901 in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 202108058MINB
Record Dates: First submitted 2021-09-23; First posted 2021-10-15 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2023-01

CONDITIONS: Covid19 Vaccine
Keywords: Covid19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderna COVID-19 vaccine (mRNA 1273) (Active Comparator): 110 participants will be randomly assigned to Moderna COVID 19
  Interventions: Biological: Homologous boost schedule
- Medigen COVID-19 vaccine (MVC COV1901) (Experimental): 110 participants will be randomly assigned to Medigen COVID 19 vaccine
  Interventions: Biological: Heterologous boost schedule

INTERVENTIONS:
Biological: Homologous boost schedule — 1st dose mRNA 1273 , 2nd dose mRNA 1273
  Arms: Moderna COVID-19 vaccine (mRNA 1273)
Biological: Heterologous boost schedule — 1st dose mRNA 1273 , 2nd dose MVC COV1901
  Arms: Medigen COVID-19 vaccine (MVC COV1901)

SUMMARY:
The primary objective of the study is to evaluable the safety and to demonstrate the immunogenicity of heterologous prime-boost (mRNA-1273, MVC-COV1901), compared to homologous prime-boost (mRNA-1273), with an interval of 8-12 weeks, This study also assesses the safety and tolerability of the study intervention and explores the immunogenicity by the antigen-specific immunoglobulin, the immunogenicity against the VoCs, the antigen specific cellular immune response, as well as the potential efficacy of study intervention in preventing COVID-19.

DETAILED DESCRIPTION:
This is a parallel group, prospective, randomized, double-blind, two-arm, single-center study to be conducted in approximately 220 healthy participants aged 20 to 70 years who are generally healthy or with stable pre-existing health condition.

The participants should previously have their first dose of mRNA-1273. The participants, investigators, and the site personnel will be blinded to the study intervention assignment until all the participants complete their Day 29. Preparation and administration of study intervention will be performed by authorized unblinded site personnel who do not participate in the evaluation of the participants.

Eligible participants will be randomized to receive either mRNA-1273 or MVC-COV1901 vaccine at a 1:1 ratio. Randomization of participants will be stratified by the interval apart from their first dose of mRNA-1273 (< 10 weeks or ≥ 10 weeks).

The study consists of 6 on-site visits:

Day -28 to Day 1, Visit 1 (Screening) Day 1, Visit 2 (study intervention) Day 15 ± 3 days, Visit 3 Day 29 ± 3 days, Visit 4 Day 91 ± 14 days, Visit 5 Day 181 ± 14 days, Visit 6 Unscheduled visit(s) may be arranged when deemed necessary by the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participant aged ≥20 to <70 years at randomization.
2. Has received one dose of the mRNA-1273 8 to 12 weeks before randomization.
3. Female participant must:

   1. Be either of non-childbearing potential, i.e. surgically sterilized (defined as having undergone hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy; tubal ligation alone is not considered sufficient) or one year post-menopausal;
   2. Or, if of childbearing potential, be abstinent or agree to use medically effective contraception from 14 days before screening to 30 days following the last administration of study intervention. Acceptable forms include:

   i. Implanted hormonal methods of contraception or placement of an intrauterine device or intrauterine system ii. Established use of hormonal methods (injectable, pill, patch or ring) combined with barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository c. Have a negative pregnancy test
4. Participant is willing and able to comply with all required study visits and follow-up required by this protocol.
5. Participant or the participant's legal representative must understand the procedures of the study and provide written informed consent.

Exclusion Criteria:

1. Pregnant or breast feeding or have plan to become pregnant within 30 days after the administration of study intervention.
2. Currently receiving or received any investigational intervention within 30 days prior to the study intervention.
3. Administered any licensed live-attenuated vaccines within 28 days or other licensed non-live-attenuated vaccines within 7 days prior to the study intervention.
4. Administered any blood product or intravenous immunoglobulin administration within 12 weeks prior to the study intervention.
5. Currently receiving or anticipate to receive concomitant immunosuppressive or immune-modifying therapy (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or < 2 weeks of daily receipt of prednisone less than 20 mg or equivalent) within 12 weeks prior to the study intervention.
6. Currently receiving or anticipate to receive treatment with tumor necrosis factor (TNF)-α inhibitors, e.g. infliximab, adalimumab, etanercept within 12 weeks prior to the study intervention.
7. Major surgery or any radiation therapy within 12 weeks prior to the study intervention.
8. Has received any investigational or licensed COVID-19 vaccine other than mRNA-1273, or ≥ two doses of mRNA-1273.
9. Immunosuppressive illness or immunodeficient state, including hematologic malignancy, history of solid organ, bone marrow transplantation, or asplenia.
10. A history of malignancy with potential risk for recurrence after curative treatment, or current diagnosis of or treatment for cancer (exceptions are squamous and basal cell carcinomas of the skin and treated uterine cervical carcinoma in situ, at the discretion of the investigator).
11. Bleeding disorder considered a contraindication to IM injection or phlebotomy.
12. Known SARS-CoV-2 infection in the recent 3 months prior to the study intervention.
13. A history of cerebral venous sinus thrombosis, heparin-induced thrombocytopenia or antiphospholipid syndrome.
14. Participant who, in the investigator's judgement, is not in a stable condition and by participating in the study could adversely affect the safety of the participant, interfere with adherence to study requirements or evaluation of any study endpoint. This may include a participant with ongoing acute diseases, severe infections, autoimmune disease, laboratory abnormality or serious medical conditions in the following systems: cardiovascular, pulmonary, hepatic, neurologic, metabolic, renal, or psychiatric.
15. A history of hypersensitivity to any vaccine or a history of allergic disease or reactions likely to be exacerbated by any component of the mRNA-1273 or MVC-COV1901.
16. Body (oral, rectal, or ear) temperature ≥ 38.0°C or acute illness (not including minor illnesses such as diarrhea or mild upper respiratory tract infection at the discretion of the investigator) within 2 days before the study intervention.

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Primary Immunogenicity-GMT | Day 1 to Day 15
  To evaluate the immunogenicity of heterologous prime boost (mRNA 1273, MVC-COV1901), compared to homologous prime boost (mRNA 1273), in terms of neutralizing antibody titers at 14 days after the study intervention
  -Geometric mean titer (GMT)
Primary Immunogenicity-SCR | Day 1 to Day 15
  To evaluate the immunogenicity of heterologous prime boost (mRNA 1273, MVC-COV1901), compared to homologous prime boost (mRNA 1273), in terms of neutralizing antibody titers at 14 days after the study intervention
  -Seroconversion rate (SCR)
Primary Immunogenicity-GMR | Day 1 to Day 15
  To evaluate the immunogenicity of heterologous prime boost (mRNA 1273, MVC-COV1901), compared to homologous prime boost (mRNA 1273), in terms of neutralizing antibody titers at 14 days after the study intervention
  -GMT ratio
Primary Safety | Day 1 to Day 29
  To evaluate the safety and tolerability of heterologous prime boost (mRNA 1273, MVC-COV1901), compared to homologous prime boost (mRNA 1273) from Day 1 to Day 29
  The number and percentage of participants with the occurrence of:
  * Solicited local adverse events (AEs)
  * Solicited systemic AEs
  * Unsolicited AEs

SECONDARY OUTCOMES:
Secondary Immunogenicity-GMT | Day 29 to Day 181
  To evaluate the immunogenicity of heterologous prime-boost (mRNA-1273, MVC-COV1901), compared to homologous prime-boost (mRNA-1273) in terms of neutralizing antibody titers at 28 days, 90 days, and 180 days after the study intervention
  -Geometric mean titer (GMT)
Secondary Immunogenicity-SCR | Day 29 to Day 181
  To evaluate the immunogenicity of heterologous prime-boost (mRNA-1273, MVC-COV1901), compared to homologous prime-boost (mRNA-1273) in terms of neutralizing antibody titers at 28 days, 90 days, and 180 days after the study intervention
  -Seroconversion rate (SCR)
Secondary Immunogenicity-GMR | Day 29 to Day 181
  To evaluate the immunogenicity of heterologous prime-boost (mRNA-1273, MVC-COV1901), compared to homologous prime-boost (mRNA-1273) in terms of neutralizing antibody titers at 28 days, 90 days, and 180 days after the study intervention
  -GMT ratio
Secondary Safety | Day 1 to Day 181
  To evaluate the safety of heterologous prime-boost (mRNA-1273, MVC-COV1901), compared to homologous prime-boost (mRNA-1273) throughout the study
  The number and percentage of participants with the occurrence of:
  * Medically Attended Adverse Events (MAAEs)
  * Adverse Event of Special Interest (AESIs)
  * Vaccine-Associated Enhanced Disease (VAED)
  * Serious Adverse Events(SAEs)

OTHER OUTCOMES:
Exploratory (antigen-specific immunoglobulin)-GMT | Day 29 to Day 181
  To evaluate the immunogenicity of heterologous prime-boost (mRNA-1273, MVC-COV1901), compared to homologous prime-boost (mRNA-1273), in terms of antigen-specific immunoglobulin titers at 28 days, 90 days, and 180 days after the study intervention
  -Geometric mean titer (GMT)
Exploratory (antigen-specific immunoglobulin)-SCR | Day 29 to Day 181
  To evaluate the immunogenicity of heterologous prime-boost (mRNA-1273, MVC-COV1901), compared to homologous prime-boost (mRNA-1273), in terms of antigen-specific immunoglobulin titers at 28 days, 90 days, and 180 days after the study intervention
  -Seroconversion rate (SCR)
Exploratory (antigen-specific immunoglobulin)-GMR | Day 29 to Day 181
  To evaluate the immunogenicity of heterologous prime-boost (mRNA-1273, MVC-COV1901), compared to homologous prime-boost (mRNA-1273), in terms of antigen-specific immunoglobulin titers at 28 days, 90 days, and 180 days after the study intervention
  -GMT ratio
Exploratory (VoC) | Day 1 to Day 15
  To evaluate the immunogenicity of heterologous prime-boost (mRNA-1273, MVC-COV1901), compared to homologous prime-boost (mRNA-1273), in terms of neutralizing antibody titers against Variants of Concerns at 14 days after the study intervention
  * GMT against VoCs including the Delta strain
  * Fold-reduction of GMT against VoCs comparing to Wild-Type strain
Exploratory (Cell Immunity) | Day 1 to Day 15
  To evaluate antigen specific cellular immune responsese of heterologous prime-boost (mRNA-1273, MVC-COV1901), compared to homologous prime-boost (mRNA-1273) at 14 days after the study intervention as determined by various classes of cytokines
Exploratory (Clinical Efficacy) | Day 15 to Day 181
  To estimate the efficacy of heterologous prime-boost (mRNA-1273, MVC-COV1901), compared to homologous prime-boost (mRNA-1273), in the prevention of COVID-19
  * Number of laboratory-confirmed COVID-19 cases occurring ≥ 15 days after study intervention
  * Number of laboratory-confirmed COVID-19 severe cases occurring ≥ 15 days after study intervention

CONTACTS AND LOCATIONS:
Overall Officials: Szu-Min Hsieh, MD.Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang ST, Huang YS, Liu WD, Pan SC, Sun HY, Lien CE, Chen C, Hsieh SM. Immunogenicity and safety of heterologous mRNA-1273/MVC-COV1901 vaccination versus homologous mRNA1273 vaccination: A randomized, double-blind controlled study. J Formos Med Assoc. 2023 Nov;122(11):1165-1173. doi: 10.1016/j.jfma.2023.05.030. Epub 2023 Jun 14. PMID 37321955